CLINICAL TRIAL: NCT00813891
Title: Efficacy of Ranibizumab (Lucentis) in Combination With Photodynamic Therapy for Neovascular Age-Related Macular Degeneration
Brief Title: Efficacy of Ranibizumab in Combination With Photodynamic Therapy for Wet Age-Related Macular Degeneration
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: McGill University Health Center, McGill Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUHC - 1234 - RVH
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Macular Degeneration; Visual Acuity
Keywords: ranibizumab; verteporfin
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pre-PDT (Active Comparator): Participants in this group will receive an intraocular Ranibizumab injection one week prior to the first PDT with verteporfin.
  Interventions: Drug: Ranibizumab
- Post-PDT (Active Comparator): Participants in this group will receive an intraocular Ranibizumab injection one week post the first PDT with verteporfin.
  Interventions: Drug: Ranibizumab
- No PDT (Active Comparator): Participants in this group will receive an intraocular Ranibizumab injection with no accompanying PDT with verteporfin.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intraocular injection of 0.5mg of Ranibizumab one week prior to PDT with verteporfin
  Other Names: Lucentis the brand name of Ranibizumab
  Arms: Pre-PDT
Drug: Ranibizumab — Intraocular injection of 0.5mg of Ranibizumab one week after PDT with verteporfin
  Other Names: Lucentis the brand name of Ranibizumab
  Arms: Post-PDT
Drug: Ranibizumab — Intraocular injection of 0.5mg of Ranibizumab with no accompanying PDT with verteporfin
  Other Names: Lucentis the brand name of Ranibizumab
  Arms: No PDT

SUMMARY:
The purpose of the investigators study is to look at the visual outcomes of Ranibizumab injections in combination with photodynamic therapy for the treatment of neovascular age-related macular degeneration.

DETAILED DESCRIPTION:
The main cause of severe vision loss in patients with age-related macular degeneration (AMD) is the development of choroidal neovascularization (CNV). This debilitating form of AMD affects the macula lutea, the central part of the retina, which is responsible for high resolution visual acuity. Characteristic findings in neovascular AMD include the development of new, abnormal blood vessels in the choroid layer beneath the macula otherwise known as CNV.

Current treatment options for this condition have included include laser therapy, photodynamic therapy (PDT), and intraocular injections (different types of anti-vascular endothelial growth factors) alone or in combination. While current treatments were demonstrated to slow the progression of vision loss, neither therapy was shown to significantly improve visual acuity.

Given their different modes of action, it is believed that combination therapy of Ranibizumab with PDT may lead to better visual outcomes and may result in an improved effect in treating AMD and therefore may help decrease the need for monthly Ranibizumab injections. After the first injection, regardless of which group the patient has been assigned to, they will receive Ranibizumab injections at 4 week intervals if clinically indicated. The purpose of the this study is to evaluate the visual outcomes of intraocular Ranibizumab injections in combination with photodynamic therapy with verteporfin for the treatment of neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with any subtype of primary subfoveal or juxtafoveal choroidal neovascularization
* must be 50 years of age or older
* have a lesion whose total size is no more than 5400micrometres in greatest linear dimension in the study eye
* CNV that is more than 50% obscured by blood
* have best corrected visual acuity of 20/50-20/320 (Snellen equivalent)
* have been assessed with the use of early treatment diabetic retinopathy study charts

Exclusion Criteria:

* previous treatment (including verteporfin therapy) that could compromise an assessment of the study treatment
* any permanent structural damage to the central fovea

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline at 6 months in the best corrected visual acuity (VA) score using an early treatment diabetic retinopathy study eye chart at a starting distance of 4 meters. | Monthly for a total of 12 months

SECONDARY OUTCOMES:
To determine the following: 1:Proportion of subjects who loose fewer than 15 letters from baseline visual acuity at 6 months 2: Proportion of subjects with VA of 20/200 or worse 3: Proportion of subjects with VA of 20/40 or better | One year

CONTACTS AND LOCATIONS:
Overall Officials: John Galic, MD, Principal Investigator — Montreal Retina Institute; John Chen, MD, Principal Investigator — Montreal Retina Institute
Locations (1):
- The Royal Victoria Hospital and the Montreal Retinal Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Bressler NM, Bressler SB, Congdon NG, Ferris FL 3rd, Friedman DS, Klein R, Lindblad AS, Milton RC, Seddon JM; Age-Related Eye Disease Study Research Group. Potential public health impact of Age-Related Eye Disease Study results: AREDS report no. 11. Arch Ophthalmol. 2003 Nov;121(11):1621-4. doi: 10.1001/archopht.121.11.1621. PMID 14609922
- [Background] Klein R, Peto T, Bird A, Vannewkirk MR. The epidemiology of age-related macular degeneration. Am J Ophthalmol. 2004 Mar;137(3):486-95. doi: 10.1016/j.ajo.2003.11.069. PMID 15013873
- [Background] Congdon N, O'Colmain B, Klaver CC, Klein R, Munoz B, Friedman DS, Kempen J, Taylor HR, Mitchell P; Eye Diseases Prevalence Research Group. Causes and prevalence of visual impairment among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):477-85. doi: 10.1001/archopht.122.4.477. PMID 15078664
- [Background] Friedman DS, O'Colmain BJ, Munoz B, Tomany SC, McCarty C, de Jong PT, Nemesure B, Mitchell P, Kempen J; Eye Diseases Prevalence Research Group. Prevalence of age-related macular degeneration in the United States. Arch Ophthalmol. 2004 Apr;122(4):564-72. doi: 10.1001/archopht.122.4.564. PMID 15078675
- [Background] Bressler NM. Age-related macular degeneration is the leading cause of blindness.. JAMA. 2004 Apr 21;291(15):1900-1. doi: 10.1001/jama.291.15.1900. No abstract available. PMID 15108691
- [Background] Resnikoff S, Pascolini D, Etya'ale D, Kocur I, Pararajasegaram R, Pokharel GP, Mariotti SP. Global data on visual impairment in the year 2002. Bull World Health Organ. 2004 Nov;82(11):844-51. Epub 2004 Dec 14. PMID 15640920
- [Background] Yannuzzi LA, Negrao S, Iida T, Carvalho C, Rodriguez-Coleman H, Slakter J, Freund KB, Sorenson J, Orlock D, Borodoker N. Retinal angiomatous proliferation in age-related macular degeneration. Retina. 2001;21(5):416-34. doi: 10.1097/00006982-200110000-00003. PMID 11642370
- [Background] Holz FG, Pauleikhoff D, Klein R, Bird AC. Pathogenesis of lesions in late age-related macular disease. Am J Ophthalmol. 2004 Mar;137(3):504-10. doi: 10.1016/j.ajo.2003.11.026. PMID 15013875
- [Background] Lopez PF, Sippy BD, Lambert HM, Thach AB, Hinton DR. Transdifferentiated retinal pigment epithelial cells are immunoreactive for vascular endothelial growth factor in surgically excised age-related macular degeneration-related choroidal neovascular membranes. Invest Ophthalmol Vis Sci. 1996 Apr;37(5):855-68. PMID 8603870
- [Background] Frank RN, Amin RH, Eliott D, Puklin JE, Abrams GW. Basic fibroblast growth factor and vascular endothelial growth factor are present in epiretinal and choroidal neovascular membranes. Am J Ophthalmol. 1996 Sep;122(3):393-403. doi: 10.1016/s0002-9394(14)72066-5. PMID 8794712
- [Background] Kvanta A, Algvere PV, Berglin L, Seregard S. Subfoveal fibrovascular membranes in age-related macular degeneration express vascular endothelial growth factor. Invest Ophthalmol Vis Sci. 1996 Aug;37(9):1929-34. PMID 8759365
- [Background] Kliffen M, Sharma HS, Mooy CM, Kerkvliet S, de Jong PT. Increased expression of angiogenic growth factors in age-related maculopathy. Br J Ophthalmol. 1997 Feb;81(2):154-62. doi: 10.1136/bjo.81.2.154. PMID 9059252
- [Background] Otani A, Takagi H, Oh H, Koyama S, Ogura Y, Matumura M, Honda Y. Vascular endothelial growth factor family and receptor expression in human choroidal neovascular membranes. Microvasc Res. 2002 Jul;64(1):162-9. doi: 10.1006/mvre.2002.2407. No abstract available. PMID 12074642
- [Background] Rakic JM, Lambert V, Devy L, Luttun A, Carmeliet P, Claes C, Nguyen L, Foidart JM, Noel A, Munaut C. Placental growth factor, a member of the VEGF family, contributes to the development of choroidal neovascularization. Invest Ophthalmol Vis Sci. 2003 Jul;44(7):3186-93. doi: 10.1167/iovs.02-1092. PMID 12824270
- [Background] Okamoto N, Tobe T, Hackett SF, Ozaki H, Vinores MA, LaRochelle W, Zack DJ, Campochiaro PA. Transgenic mice with increased expression of vascular endothelial growth factor in the retina: a new model of intraretinal and subretinal neovascularization. Am J Pathol. 1997 Jul;151(1):281-91. PMID 9212753
- [Background] Schwesinger C, Yee C, Rohan RM, Joussen AM, Fernandez A, Meyer TN, Poulaki V, Ma JJ, Redmond TM, Liu S, Adamis AP, D'Amato RJ. Intrachoroidal neovascularization in transgenic mice overexpressing vascular endothelial growth factor in the retinal pigment epithelium. Am J Pathol. 2001 Mar;158(3):1161-72. doi: 10.1016/S0002-9440(10)64063-1. PMID 11238064
- [Background] Krzystolik MG, Afshari MA, Adamis AP, Gaudreault J, Gragoudas ES, Michaud NA, Li W, Connolly E, O'Neill CA, Miller JW. Prevention of experimental choroidal neovascularization with intravitreal anti-vascular endothelial growth factor antibody fragment. Arch Ophthalmol. 2002 Mar;120(3):338-46. doi: 10.1001/archopht.120.3.338. PMID 11879138
- [Background] Saishin Y, Saishin Y, Takahashi K, Lima e Silva R, Hylton D, Rudge JS, Wiegand SJ, Campochiaro PA. VEGF-TRAP(R1R2) suppresses choroidal neovascularization and VEGF-induced breakdown of the blood-retinal barrier. J Cell Physiol. 2003 May;195(2):241-8. doi: 10.1002/jcp.10246. PMID 12652651
- [Background] Verteporfin Roundtable 2000 and 2001 Participants; Treatment of age-related macular degeneration with photodynamic therapy (TAP) study group principal investigators; Verteporfin in photodynamic therapy (VIP) study group principal investigators. Guidelines for using verteporfin (visudyne) in photodynamic therapy to treat choroidal neovascularization due to age-related macular degeneration and other causes. Retina. 2002 Feb;22(1):6-18. doi: 10.1097/00006982-200202000-00003. PMID 11884872
- [Result] Gragoudas ES, Adamis AP, Cunningham ET Jr, Feinsod M, Guyer DR; VEGF Inhibition Study in Ocular Neovascularization Clinical Trial Group. Pegaptanib for neovascular age-related macular degeneration. N Engl J Med. 2004 Dec 30;351(27):2805-16. doi: 10.1056/NEJMoa042760. PMID 15625332
- [Result] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Result] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319